CLINICAL TRIAL: NCT00820014
Title: Evaluation of Tolerability, Safety and Ocular Pharmacokinetics of Topically Applied ESBA105 in Patients Undergoing Cataract Surgery or Combined Cataract Surgery and Vitrectomy
Brief Title: Ocular Biodistribution Study for Topically Applied ESBA105
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ESBATech AG (Industry)
Responsible Party: Peter Lichtlen, Medical Director, ESBATech AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: ESBA105CRD03
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2009-01

CONDITIONS: Cataract
Keywords: ESBA105; scFv antibody fragment; cataract surgery; pharmacokinetics; biodistribution; Irvine-Gass syndrome
MeSH Terms: conditions — Cataract; Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ESBA105 eye drops
  Interventions: Drug: Placebo
- 2 (Placebo Comparator): Placebo control (vehicle)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo control (vehicle) eye drops applied 4-times a day for 4 days before ocular surgery

SUMMARY:
The purpose of this study is to determine whether ESBA105, a single-chain (scFv) antibody against TNF-alpha, efficiently penetrates into the anterior chamber and the vitreous body upon topical administration to the eye.

DETAILED DESCRIPTION:
ESBA105 is a topically administered tumour necrosis factor alpha (TNF-alpha) inhibitor that has significant therapeutic potential in various inflammatory intraocular diseases. In animal experiments, ESBA105 was shown to efficiently penetrate into the inner of the eye upon topical administration, associated with very low systemic exposure. A recently completed Phase I trial with topical ESBA105 has confirmed the safety of topical administration to the human eye and the low systemic exposure using this route of administration.

This study is designed to determine the intraocular levels and the specific intraocular distribution pattern of ESBA105 following topical administration to the human eye. In addition it shall be explored whether topical administration of ESBA105 reduces intraocular inflammation following cataract surgery.

Three different dose regimens will be applied to four different patient cohorts. Three patient cohorts will be conducted in an open label design and one in a double-masked, placebo controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasian patients ≥18 years.
* Written informed consent prior to any study procedures including screening tests for eligibility.
* Patients should be in good health as determined by past medical history, physical examination, vital signs, electrocardiogram (ECG), and laboratory tests at screening.
* Ability to administer eye drops (personally or administered by another person).

Cataract patients:

* Eligible for routine, uncomplicated senile cataract surgery.

Vitrectomy patients:

* Diagnosis of epiretinal fibroplasia requiring vitrectomy and cataract surgery.

Exclusion Criteria:

* Treated glaucoma / elevated intraocular pressure (IOP) requiring therapy.
* History of chronic or recurrent intraocular inflammatory disease.
* Uncontrolled diabetes mellitus (fasting blood glucose >15 mmol/L).
* Diabetic retinopathy with history of laser photocoagulation.
* Patients with a single eye or a pinholed visual acuity (VA) 20/200 or worse measured on Snellen chart in the non-study eye.
* Iris atrophy in the eye to undergo surgery.
* Pregnant or breast-feeding women or women of childbearing potential, who with their partners refuse to use 2 reliable methods of contraception
* History of collagenosis or systemic vasculitis.
* Patients who have had ocular surgery (including laser surgery) in the study eye within 3 months or in the contralateral eye within 2 weeks prior to screening.
* Patients who have an active systemic or local (anywhere in the body) bacterial and/or viral infection.
* Positive or unclear QuantiFERON-TB Gold assay result.
* Participation in a clinical study with investigational drugs within 3 months prior to screening.
* Inability to comply with the study requirements.
* Patients with known, severely impaired hepatic function, or laboratory values reflecting inadequate hepatic function.
* Patients with pre-existing chronic renal failure defined by a calculated creatinine clearance (CrCl) of < 40 mL/min, using the Cockcroft-Gault estimate for glomerular filtration rate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determination of intraocular ESBA105 levels, local biodistribution (aqueous and vitreous humor) and intraocular pharmacokinetics upon topical administration. | Collection of respective biological matrices at occasion of ocular surgery

SECONDARY OUTCOMES:
Exploratory assessment of the anti-inflammatory potential of prophylactic, topical ESBA105 for prevention of post-surgical inflammation following cataract surgery. | 10 Days following ocular surgery
Assessment of local tolerability and safety of topical ESBA105. | up to 10 Days following ocular surgery
Assessment of systemic exposure upon topical application of ESBA105. | 1 Day following ocular surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Thiel, MD, PhD, Principal Investigator — Kantonsspital Luzern, Augenklinik, CH-6000 Luzern 16, Switzerland
Locations (2):
- Switzerland (2):
  - Kantonsspital Luzern, Augenklinik, CH-6000 Luzern 16, Switzerland, Lucerne, Canton of Lucerne
  - Pallas Gruppe, Olten, Canton of Solothurn